CLINICAL TRIAL: NCT02271607
Title: A Pilot Study About The Effects of Indirect-Moxibustion on Bladder- Functional Improvement and Symptoms Management in Patients With Overactive Bladder: A Randomized Controlled Trial
Brief Title: The Effect and Safety of Moxibustion Therapy for Overactive Bladder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Principal Investigator, JUNGNAM KWON, Professor, Korean Medicine Hospital of Pusan National University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201405
Record Dates: First submitted 2014-10-11; First posted 2014-10-22 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Overactive Bladder; Hyperthermia; Urinary Frequency or Urgency Adverse Event; Lower Urinary Tract Symptoms
Keywords: moxibustion
MeSH Terms: conditions — Urinary Bladder, Overactive; Hyperthermia; Lower Urinary Tract Symptoms | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- moxibustion (Experimental): A series of moxibustion sessions within four weeks from the baseline followed by observation period of four weeks.
  Interventions: Device: moxibustion
- waiting (No Intervention): Waiting period of four weeks followed by moxibustion therapy sessions on the same way with moxibustion group.

INTERVENTIONS:
Device: moxibustion — The treatment schedule is three times per week for four weeks. Indirect moxa pillars and indirect-container moxibustion will be used.
  Other Names: moxa pillar
  Arms: moxibustion

SUMMARY:
This pragmatic randomized controlled study aimed to evaluate the effectiveness and safety of moxibustion therapy on overactive bladder (OAB) patients.

DETAILED DESCRIPTION:
Patients who diagnosed as overactive bladder aged 20 to 75 years old will be divided into two groups, one is moxibustion-therapy and the other is waiting-list group.

Patients who belong to moxibustion therapy group will be treated moxibustion for 12 times by a Korean Medicine doctor.

Patients who belong to waiting-list group will be prohibited to get any treatment including moxibustion for relieve the symptoms of overactive bladder, and the same moxibustion therapy with moxbiustion-therapy group will be conducted after 4 weeks.

Overactive bladder symptom score (OABSS), overactive bladder-validated 8-question (OAB-V8) will be measured to evaluate the effectiveness.

The number of side effect will be measured to evaluate the safety.

The skin temperature of CV4, SP6 and LR3, and the tympanic temperature will be measured to study treatment mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. aged from 20 to 75 years old
2. submit written consent
3. no deficit to notify the hotness promptly and exactly
4. diagnosed with overactive bladder
5. suffering the OAB symptoms during greater than or equal to 3 months

Exclusion Criteria:

1. malignancy
2. obstructive disease of urinary tract
3. cystocele, vaginocele or rectocele
4. urinary tract infection finding on urine analysis
5. diabetic mellitus
6. sensory disturbance
7. pregnancy, possibility of pregnancy or planning to pregnancy
8. problems to communication due to any medical problem such as cognitive dysfunction
9. getting other treatment of either Traditional Korean Medicine or conventional medicine for overactive bladder
10. psychiatric disorder or severe systemic disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overactive bladder-validated 8-questions | 4 weeks
  This is to measure how the patients have been bothered by OAB.

SECONDARY OUTCOMES:
Overactive bladder symptom scores | 4, 8 weeks
  self-administered questionnaire about daytime frequency, nighttime frequency, urgency and urgency incontinence.
The skin temperature of CV4, SP6 and LR3 | 4, 8 weeks
  this is to establish the foundation of researching moxibustion-therapy mechanism.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Nam Kwon, PhD, Study Chair — Korean Medicine Hospital, Pusan National University
Locations (1):
- National Clinical Research Center, Korean Medicine Hospital, Pusan National University, Yangsa, Kyungsangnamdo, South Korea

REFERENCES:
- [Result] Lee MS, Choi TY, Park JE, Lee SS, Ernst E. Moxibustion for cancer care: a systematic review and meta-analysis. BMC Cancer. 2010 Apr 7;10:130. doi: 10.1186/1471-2407-10-130. PMID 20374659
- [Result] Chiu JH. How does moxibustion possibly work? Evid Based Complement Alternat Med. 2013;2013:198584. doi: 10.1155/2013/198584. Epub 2013 Mar 27. PMID 23606872
- [Result] Guo ZF, Liu Y, Hu GH, Liu H, Xu YF. Transcutaneous electrical nerve stimulation in the treatment of patients with poststroke urinary incontinence. Clin Interv Aging. 2014 May 23;9:851-6. doi: 10.2147/CIA.S61084. eCollection 2014. PMID 24904204
- [Result] Jeong SJ, Homma Y, Oh SJ. Reproducibility study of Overactive Bladder Symptom Score questionnaire and its response to treatment (RESORT) in Korean population with overactive bladder symptoms. Qual Life Res. 2014 Feb;23(1):285-92. doi: 10.1007/s11136-013-0440-7. Epub 2013 May 29. PMID 23715806
- [Result] Takeda M, Nishizawa O, Gotoh M, Yoshida M, Takahashi S, Masumori N. Clinical efficacy and safety of imidafenacin as add-on treatment for persistent overactive bladder symptoms despite alpha-blocker treatment in patients with BPH: the ADDITION study. Urology. 2013 Oct;82(4):887-93. doi: 10.1016/j.urology.2013.05.008. Epub 2013 Aug 14. PMID 23953605
- [Derived] Lee HY, Yun YJ, Choi JY, Hong JW, Lee I, Park SH, Kwon JN. Effectiveness and safety of moxibustion for alleviating symptoms of overactive bladder: A prospective, randomized controlled, crossover-design, pilot study. Medicine (Baltimore). 2018 Aug;97(34):e12016. doi: 10.1097/MD.0000000000012016. PMID 30142847